CLINICAL TRIAL: NCT06370533
Title: The Effects of Mobile Health Based Lifestyle Intervention on Gestational Weight Gain in Pregnant Women With Overweight and Obesity: A Randomized Controlled Trial
Brief Title: Healthy Gestational Weight Gain Programme
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Peking University Health Science Center-Weifang Joint Research Center for Maternal and Child Health (Unknown); W.F. Maternal and Child Health Hospital (Unknown); Tongzhou Maternal and Child Health-care Institution of Beijing (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HGWG-pro
Record Dates: First submitted 2024-03-31; First posted 2024-04-17 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-05

CONDITIONS: Gestational Weight Gain; Overweight and Obesity
MeSH Terms: conditions — Gestational Weight Gain; Overweight; Obesity | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lifestyle intervention (Experimental): Health education: Individual face to face or telephone sessions and online health education material.
  Diet behavior: The eight eating behavioral goals will be assigned to each participant with two for every 4-week cycle.
  Physical activity: Women will be advised to gradually attaining the goal of 150 minutes of moderate- to vigorous-intensity physical activity per week and walk at least 6000 steps per day.
  Weight monitoring: Self-monitoring of weight gain (regular self-weighing) and weight logging at least once a week was recommended.
  Interventions: Behavioral: behavioral interventions
- usual-care control (No Intervention): Provision of usual prenatal care

INTERVENTIONS:
Behavioral: behavioral interventions — The investigators set diet, physical activity, and weight goals for each participant. During the lifestyle intervention period, the participants need to complete weekly self-monitoring of weight, weekly recording of diet behavioral goals, timely exercise logging, online health education course learning by using the WeChat public account. They will receive corresponding timely reminder and tailored feedback in the form of graphical illustration and text according to diet, physical activity, and weight data collected by WeChat public account and Huawei Wristband. They will receive individual face to face or telephone sessions every 2 weeks to complete health education, goal review, motivational interview as well as collecting adverse events.
  Arms: lifestyle intervention

SUMMARY:
This study aims to evaluate the efficacy of a multi-component lifestyle interventions during pregnancy on promoting appropriate gestational weight gain, preventing GDM, and improving pregnancy, delivery, and neonatal outcomes among overweight or obese pregnant women. The intervention strategies are developed based on the transtheoretical model and mobile health (via WeChat Public Account in smartphone), and will be conducted online and offline. This study will recruit and follow-up 200 overweight or obese singleton pregnant women (pre-pregnancy 24kg/m2≤BMI≤40 kg/m2) during the first trimester of pregnancy from Weifang Maternal and Child Health Hospital, Shandong Province, China, and Tongzhou Maternal and Child Health-care Institution, Beijing, China, with 100 pregnancy women in each institution. The 200 overweight or obese pregnant women will be randomly allocated at a 1:1 ratio to either the intervention or control group, stratified by the categorical variables of age, BMI and parity. Participants in the control group will be provided usual prenatal care. The lifestyle intervention will last for approximately 6 months (from 10-14 weeks to 32-36 weeks of gestation). Follow-up timepoints included 8-14 weeks of gestation, 24-28 weeks of gestation, 32-36 weeks of gestation. The interventions are composed of health education related to gestational weight gain and healthy lifestyles, diet modification, active physical activity, regular individual in-person and telephone sessions, diet behavior monitoring, physical activity monitoring, and weight monitoring with Huawei Wristband and WeChat Public Account. The hypothesis is that lifestyle interventions based on the transtheoretical model and mobile health will result in more appropriate gestational weight gain and lower risk of adverse pregnancy outcomes compared with usual care.

DETAILED DESCRIPTION:
Overweight and obesity is a major public health problem among women in reproductive age. Excessive gestational weight gain (EGWG) among this group is becoming a worldwide epidemic over recent decades. EGWG is associated with adverse outcomes including increased risk of developing gestational diabetes mellitus (GDM), cesarean section, hypertensive disorders of pregnancy (HDP), elevated infant birth weight and adiposity, and increased risk of metabolic syndrome and childhood obesity in offspring. Therefore, interventions are needed to help overweight and obese pregnant women to control GWG.

Lifestyle intervention has been proved effective on weight management during pregnancy. However, the effects of interventions on controlling overweight and obese women's GWG are inconsistent. Traditional face-to-face counseling are less cost effective. Effective intervention models based on Mobile health that can be scaled up are scarce. Thus, this randomized controlled trial aims to identify: firstly, whether the mobile health lifestyle interventions will be effective on improving gestational weight gain and preventing GDM among overweight or obese pregnant women; secondly, whether the intervention will be beneficial for improving pregnancy outcomes, delivery outcomes, neonatal outcomes, metabolic indicators, body composition indicators, etc. among overweight or obese pregnant women.

The interventions are composed of health education (online and offline health education on recommended gestational weight gain, prenatal dietary guidance and physical activity recommendation), diet behavior modification (8 core dietary goal setting and monitoring weekly), active physical activity (150 min per week of moderate-to vigorous-intensity physical activity including aerobic exercise (brisk walking) and resistance exercise; goal of 6000 steps/day), regular face to face or telephone sessions, lifestyle (diet and physical activity behavior) and weight monitoring via Huawei Wristband or WeChat Public Account. Tailoring of the intervention will be guided by the transtheoretical model. A total of 200 overweight or obese singleton pregnant women of 8-14 weeks of gestation will be recruited and they will be randomly allocated at a 1:1 ratio to either the intervention or control group, stratified by the categorical variables of age, BMI and parity. Participants in the control group will be provided usual prenatal care.

Women in both study arms will attend three research appointments at 8-14 weeks (baseline),24-28 weeks (midterm) and 32-36 weeks (terminal) of gestation for data collection via questionnaires, physical measurements, and clinical laboratory examination. Information on demography, socioeconomic status, medical and family history, obstetric history, current pregnancy information, smoking, consumption of alcohol, attitude and knowledge about GWG, diet and exercise habits, sleep situation, quality of life, mental health (depression, anxiety), social support, self-efficacy, etc. will be collected with questionnaires and interviews by research stuff. Physical measurements including weight, height, blood pressure, and body composition using bioelectrical impedance (BIA) will be obtained using standardized methods. Laboratory tests performed in conjunction with antenatal visits include a 75 g 2-hour oral glucose tolerance test (OGTT). Data on mode of delivery, gestational age at birth, birth weight, Apgar scores, perinatal complications, etc. will be obtained from patient records. In addition, blood and urine samples will be drawn at three appointments and a sample of cord blood will be collected at birth. Maternal postpartum weight (42 days,6 months,1 year after delivery) will be obtained through routine physical examination or telephone follow-up. Offspring physical growth indicators, such as height, weight, head circumference, etc., will be collected from routine physical examination in 42 days, 6 months and 12 months of age.

ELIGIBILITY:
Inclusion Criteria:

1. At 8-14 weeks of gestation
2. Overweight or obese (pre-pregnancy 40 kg/m2≥BMI≥24 kg/m2) based on BMI recommendations of the Group of China Obesity Task Force of the Chinese Ministry of Health accounting for interracial differences (overweight BMI 24-28 kg/m2 and obese BMI≥28kg/m2)
3. 18-40 years of age
4. Singleton pregnant
5. Skilled at using smartphones and WeChat during pregnancy
6. Attend regular antenatal care and plan delivery at W.F. Maternal and Child Health Hospital or Tongzhou Maternal and Child Health-care Institution of Beijing
7. No contraindications to physical activity according to Physical Activity Readiness Questionnaire (PAR-Q)
8. Willing to be randomized and cooperate with research and regular follow-up visits and sign informed consent.

Exclusion Criteria:

1. Pre-pregnancy hypertension, severe cardiovascular and cerebrovascular diseases, respiratory disease, hepatic and renal disease, malignant tumors, systemic lupus erythematosus, thyroid disease, severe anemia, and other chronic consumptive diseases.
2. Cervical insufficiency (historical painless cervical dilation leading to recurrent second-trimester births in the absence of other causes; dilated cervix on manual or speculum examination, etc.), multiple pregnancy, or continuous vaginal bleeding, etc.
3. Diabetes before pregnancy
4. Special dietary needs (e.g. , vegetarianism)
5. Severe psychiatric disorders (serious mental health disorders including depression, anxiety, bipolar disorders, etc.)
6. Cognitive impairment, visual impairment or hearing impairment
7. History of bariatric surgery or surgical history involving important organs within 3 months
8. Participated in other clinical trials within 6 months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Total gestational weight gain | From pre-pregnancy to gestational week 32-36
  Weight at gestational week 32-36 minus pre-pregnancy weight (kilograms)
Gestational weight gain before OGTT screening | From pre-pregnancy to midterm (24-28 weeks)
  Gestational weight gain before OGTT screening at 24-28 weeks (kilograms)

SECONDARY OUTCOMES:
Weekly rate of gestational weight gain between study clinical assessments | Gestational weight gain from pre-pregnancy/baseline (8-14 weeks) to midterm (24-28 weeks)/terminal (32-36 weeks)
  Gestational weight gain between pre-pregnancy/baseline (8-14 weeks) and midterm (24-28 weeks)/terminal (32-36 weeks) divided by the number of weeks (kilograms per week)
Proportion of women who exceed the IOM guidelines' weekly rate of gestational weight gain between clinical assessments | From pre-pregnancy/baseline (8-14 weeks) to midterm (24-28 weeks)/terminal (32-36 weeks)
  Exceeding the weekly rate of gestational weight gain according to Institute of Medicine guidelines was defined as being above the sum of the upper limit for the first trimester (2.0 kg)+upper limit for the weekly rate (0.33 kg for overweight, 0.27 kg for obesity) ×number of weeks in the second and/or third trimesters (ie, up until the last measured pregnancy weight).
Rate of Gestational Diabetes Mellitus diagnosed according to International Association of Diabetes and Pregnancy Study Group (IADPSG) criteria | OGTT screening at 24-28 gestational weeks
  Fasting plasma glucose (FPG) ≥ 5.1 mmol/L, and/or 1-h blood glucose ≥ 10.0 mmol/L, and/or 2-h blood glucose ≥ 8.5 mmol/L
Rate of Preeclampsia/Gestational hypertension | From 20 weeks of gestation to delivery
  Preeclampsia was defined according to the criteria of the American College of Obstetricians and Gynecologists (ACOG) i.e. systolic blood pressure of ≥ 140 mmHg or diastolic blood pressure of ≥ 90 mmHg occurring after 20 weeks of gestation in a previously normotensive woman combined with new-onset proteinuria of ≥0.3 g/24 h. Gestational hypertension was defined similarly but without the presence of proteinuria.
Rate of Cesarean Section | At delivery
  Cesarean Section
Absolute/Mean Infant birth weight | At delivery
  Birth weight at delivery（kilograms）
Rate of Macrosomia | At delivery
  Infant birth weight of ≥ 4000g
Absolute/Mean Apgar scores at 1 min or 5 min | At delivery
  Apgar scores at 1 min or 5 min evaluates the baby's heart rate, respiratory effort, muscle tone, reflex irritability, and color. Each category is scored from 0 to 2, and the total score ranges from 0 to 10. A higher Apgar score indicates that the newborn is in good health.

OTHER OUTCOMES:
Change of Blood pressure | From baseline (8-14 weeks) to midterm (24-28 weeks)/terminal (32-36 weeks)
  Systolic blood pressure and diastolic blood pressure (mmHg) will be measured by using electronic sphygmomanometer
Change of body fat percentage (%) | From baseline (8-14 weeks) to midterm (24-28 weeks)/terminal (32-36 weeks)
  measure body fat percentage by bioelectrical impedance analysis
Change of fat free mass (kg) | From baseline (8-14 weeks) to midterm (24-28 weeks)/terminal (32-36 weeks)
  measure body fat free mass by bioelectrical impedance analysis
Change of muscle mass (kg) | From baseline (8-14 weeks) to midterm (24-28 weeks)/terminal (32-36 weeks)
  measure muscle mass by bioelectrical impedance analysis
Change of Attitude and knowledge | From baseline (8-14 weeks) to midterm (24-28 weeks)/terminal (32-36 weeks)
  Attitude and knowledge about gestational weight gain and weight management measured by 8 questions: ①Perceived weight category; ②The importance of knowing the recommended weight gain during pregnancy ③The best amount of weight to gain in pregnancy ④The harm of too much weight gain in pregnancy for the mother ⑤The harm of too much weight gain in pregnancy for the baby ⑥Whether the energy needs vary according to the early, middle and late stages of pregnancy ⑦Is it right to eat for two during pregnancy? ⑧Ways to manage weight gain in pregnancy According to each question pregnant women answer the correct or not to score, answer the correct for 1 point, error for 0, the total score ranged form 0 to 8 points. The higher the score the more healthy attitude and knowledge
Change of dietary intake | From baseline (8-14 weeks) to midterm (24-28 weeks)/terminal (32-36 weeks)
  Dietary intake measured by food frequency questionnaire (FFQ) investigating the frequency of food consumption over the past one month. The dietary balance index for pregnancy will be obtained according to whether the food intake of pregnant women reached the Chinese standard for pregnant women. The dietary balance index for pregnancy includes low bound score (-60 to 0), high bound score (0 to 44) and dietary quality distance (-60 to 44). The closer these three scores get to 0, the healthier the pregnant woman's diet.
Change of physical activity | From baseline (8-14 weeks) to midterm (24-28 weeks)/terminal (32-36 weeks)
  Physical activity will be measured by International Physical Activity Questionnaire-Short Form (IPAQ-SF). It asks about the frequency and duration of various types of physical activities over the past 7 days. The metabolic equivalent (MET) for different types of activities will be calculated as below and the higher score means the higher physical activity level:
  walking MET-minutes/week = 3.3 × walking minutes × walking days; moderate MET-minutes/week = 4.0 × moderate-intensity activity minutes × moderate-intensity activity days; vigorous MET-minutes/week = 8.0 × vigorous-intensity activity minutes × vigorous-intensity activity days; total physical activity MET-minutes/week = walking + moderate + vigorous MET-minutes/week.
Change of sleep quality | From baseline (8-14 weeks) to midterm (24-28 weeks)/terminal (32-36 weeks)
  Sleep quality will be measured by Pittsburgh Sleep Quality Index (PSQI). The score ranges from 0 to 21 and the higher score indicates the higher sleep quality.
Change of Quality of life (12-Item Short Form Survey, SF-12) | From baseline (8-14 weeks) to midterm (24-28 weeks)/terminal (32-36 weeks)
  Quality of life will be measured by 12-Item Short Form Survey (SF-12). The score ranges from 0 to 100 and the higher score indicates the higher quality of life.
Incidence of depression | From baseline (8-14 weeks) to midterm (24-28 weeks)/terminal (32-36 weeks)
  Depression will be measured by 9-item Patient Health Questionnaire (PHQ-9). The score ranges from 0 to 27 and the higher score indicates higher level of depression. A score greater than 4 indicates depression.
Incidence of anxiety | From baseline (8-14 weeks) to midterm (24-28 weeks)/terminal (32-36 weeks)
  Anxiety will be measured by Zung's Self Rating Anxiety Scale (SAS). The score ranges from 25 to 100 and the higher score indicates higher level of anxiety. A score greater than 49 indicates anxiety.
The Change of Self-efficacy score (General Self-Efficacy Scale, GSES) | From baseline (8-14 weeks) to midterm (24-28 weeks)/terminal (32-36 weeks)
  Self-efficacy will be measured by General Self-Efficacy Scale (GSES). The score ranged from 10 to 40 and the higher score indicates higher level of self-efficacy.
The stage of change related to gestational weight control behavior | From baseline (8-14 weeks) to midterm (24-28 weeks)/terminal (32-36 weeks)
  The investigators will use two items to assess it. "Have the participants started to adjust their diet/physical activity to control their weight during pregnancy?", "No and I do not plan to do so in the next 6 months/No, but I am ready to start within the next 6 months/No, but I am ready to start in the next 30 days/Yes, but not regularly/Yes, I am currently controlling my weight by adjusting my diet/physical activity regularly, but it has not reached 6 months /Yes, I have been controlling my weight for more than 6 months by adjusting my diet/physical activity" choices will be provided.
Rate of Postpartum weight retention | 42 days, 6 months, 1 year after delivery
  Maternal postpartum weight will be obtained through routine physical examination or telephone follow-up.
Absolute/mean offspring weight in kilograms | 42 days, 6 months and 1 year after birth.
  The difference between arms in offspring's weight.
Absolute/mean offspring height in centimetres | 42 days, 6 months and 1 year after birth.
  The difference between arms in offspring's height.
Absolute/mean offspring head circumference | 42 days, 6 months and 1 year after birth.
  The difference between arms in offspring's head circumference.

CONTACTS AND LOCATIONS:
Overall Officials: Haixue Wang, Doctor, Principal Investigator — Peking University
Locations (2):
- China (2):
  - Tongzhou Maternal and Child Health-care Institution, Beijing, Beijing Municipality
  - W.F. Maternal and Child Health Hospital；, Weifang, Shandong

IPD SHARING:
Plan to Share IPD: No